CLINICAL TRIAL: NCT04479670
Title: Psychometric and Patholinguistic Assessment of Psychotrauma Related to Natural Hazards in the Commune of "Le Prêcheur"
Acronym: EP3LAN
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Centre de recherche en Épidémiologie et Santé des Populations (CESP) (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); SOS KRIZ (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19_RIPH3-20
Record Dates: First submitted 2020-07-10; First posted 2020-07-21 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Psychological Trauma; Posttraumatic Stress Disorder PTSD; Mass Casualty Incidents
Keywords: Psychometrics; Patholinguistics; Psychotraumatism; Posttraumatic Stress Disorder PTSD; Natural hazard; Crisis management
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project is to study the evolution of mental health in a little town of the French Martinique (Le Prêcheur) by using an innovative method of analysis that combines patholinguistic and psychometric indications for patients who risk of developing psychotrauma due to a natural hazard. Investigators will gather precise and factual data concerning the psychic and mental state of the population, by collecting patients' feelings and sentiments through individual interviews and audio recordings that will be then transcribed, and analyzed, and repeated, according to a quantitative, qualitative, and prospective methodology.

This research is launched in order to meet the needs expressed both by the French authorities and the population towards an optimization of crisis management.

DETAILED DESCRIPTION:
The study focuses on the town of Le Prêcheur (1600 inhabitants) which has a geographical location of dangerous threat at the foot of the Pelee volcano, generating intense stress and psychotraumatic disorders. Indeed, faced with the phenomena of mudslides and boulders in connection with volcanic activity (Lahars) and repeated alerts, several cases of Psychotrauma have already been reported. Even if the municipal, territorial and state authorities have put in place a large-scale action to keep the population safe, the process of moving the neuralgic centers of the town will not be completed until 2021.

In the meantime, investigators propose to provide appropriate support for this situation via the SOS Kriz platform and the Psychotraumatology center of Martinique University Hospital.

In order to reach this objective, the study team will conduct patholinguistic procedures to the verbal recordings of persons from the town of Le Prêcheur every six months during one year. This analysis is carried out semi-automatically using a cognitive-discursive analysis software (Tropes1).

Two validated psychometric tests (GHQ-12 and PCL-5) to supplement the patholinguistic data will be used.

This mixed trial aims to evaluate the evolution of the overall state of mental health of the population via a patholinguistic and psychometric measurement device, to be able to target the actions of care and support to victims of psychotrauma related to risks of natural disaster in the commune of Prêcheur in Martinique.

ELIGIBILITY:
Inclusion Criteria:

* Individual over 18,
* Residing on the town of Le Prêcheur,
* Having been informed of the study,
* And having made a non-opposition decision to participate in the study.

Exclusion Criteria:

* Individual under the protection of justice or under guardianship,
* Individual with cognitive impairment incompatible with the collection of information,
* Individual who has undergone head trauma for less than one year or with residual clinical symptoms of trauma regardless of seniority,
* Individual with a proven serious suicidal risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults subjects living in the commune of "Le Prêcheur" in Martinique
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Word frequency calculation | 12 months
  The software calculates word frequency used in transcripts, drawing on their number of occurrences and grouping them by linguistic category (modalisation, verb, noun, adjective, pronoun, negation, etc.).
  Objective: define keywords according to their frequency.
  Expected Result: List of categories of words present in the speech with indication of a frequency percentage for each category as well as list of the most popular categories frequent.
Repository classification of words | 12 months
  The software groups the most frequent words in "reference universes", relying on their proximity or distance by relation to a key word which represents a central concept (e.g. feeling, feeling, behavior, time, family, crisis, etc.).
  Objective: Group the most frequent words by semantic affinities.
  Expected result: List of keywords in each reference universe.
Patholinguistic classification of words | 12 months
  The expert analyst intervenes to relate the key words of the discourse to definitive concepts of the targeted pathologies (ex. reviviscence, avoidance, negativity, reactivity, etc.).
  Objective: Constitute a predictive scenario concerning the pathology.
  Expected result: A reference table of patholinguistic concepts.
Visualization of reference universes | 12 months
  The software presents the keywords under form of concentric circles representing the semantic fields, indicating both the weight of each word (by varying the size of the circle) and its proximity or distance compared to the other keywords (on the different rings).
  Objective: Obtain a cognitive and mental representation of the speech.
  Expected result: Image representing the center and the periphery of a reference universe.
Application of the patholinguistic scenario | 12 months
  The analyst applies to the general reference universe, statically defined by the software, its specific reading grid (the patholinguistic scenario).
  Objective: Obtain a patholinguistic representation of the speech.
  Expected result: Image representing the center and the periphery of a patholinguistic concept

SECONDARY OUTCOMES:
Assess the overall mental health status | 12 months
  The corresponding score for each subject will be used to answer the General Health Questionnaire in 12 items, for the overall measure of mental health.
  The minimum value is 0, the maximum value is 12. A score greater than or equal to 2 would correspond to a psychiatric disorder.
  The difference for each subject between the GHQ-12 score at inclusion and patholinguistic quantitative variables collected at inclusion M0 and repeated at M6 and M12.
Evaluate the symptomatology of psychotrauma patients | 12 months
  The Posttraumatic Stress Disorder CheckList Scale in 20 items will be used for screening and monitoring PTSD.
  The minimum value is 0, the maximum value is 80. A threshold value of 38 suggests the presence of PTSD.
  The difference for each subject between the PCL-5 score at inclusion and patholinguistic quantitative variables collected at inclusion M0 and repeated at M6 and M12.

CONTACTS AND LOCATIONS:
Overall Officials: Louis JEHEL, PhD, Principal Investigator — CHU de Martinique
Locations (1):
- CHU of Martinique, Fort-de-France, Martinique